CLINICAL TRIAL: NCT02139748
Title: The Clinical Effect of Implant Placement and Simultaneous Grafting Using Acellular Dermal Matrix Allograft vs. Acellular Dermal Matrix Allograft Plus Bovine-Derived Xenograft
Brief Title: The Clinical Effect of Implant Placement With a Simultaneous Soft Tissue Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, DMD, MSD, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14.0387
Record Dates: First submitted 2014-04-25; First posted 2014-05-15 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2014-05

CONDITIONS: Dental Implants
Keywords: Dental Implants; Alveolar Bone Grafting; Acellular Dermis
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dental Implant & ADM (Active Comparator): Dental implant placement plus simultaneous grafting use one layer of ADM.
  Interventions: Procedure: Dental Implant & ADM
- Dental Implant & ADM & bone xenograft (Experimental): Dental implant placement plus simultaneous grafting use one layer of ADM with bovine xenograft.
  Interventions: Procedure: Dental Implant & ADM; Procedure: Dental Implant & ADM & bone xenograft

INTERVENTIONS:
Procedure: Dental Implant & ADM — A dental implant will be placed and the buccal soft tissue will be grafted using an acellular dermal matrix allograft.
Procedure: Dental Implant & ADM & bone xenograft — A dental implant will be placed along with a buccal acellular dermal matrix allograft which will cover a bone xenograft.
  Arms: Dental Implant & ADM & bone xenograft

SUMMARY:
Dental implant placement and simultaneous grafting using one layer gum graft will result in the same facial ridge contour and soft tissue thickness as one layer of gum graft plus bone graft.

DETAILED DESCRIPTION:
30 patients will have a dental implant placed in maxillary sites from teeth number 4 to 13. Any implant system is acceptable since the objective of the study is to evaluate soft tissue thickness due to graft placement, not to evaluate the implant. 15 patients will be randomly selected by a coin toss to receive a one layer of ADM (Control Group) while another fifteen will receive one layer of ADM and bovine-derived xenograft (Test Group). The graft will be placed simultaneously with the dental implant. A blinded examiner will be used. Should the examiner become unblinded the subject will be excluded from the study.

Each patient will receive a diagnostic work-up including standardized radiographs (periapicals), study casts, clinical photographs, and a periodontal examination. Presurgical preparation will include detailed oral hygiene instructions. Baseline data will be collected at initial exam. Parameters measured will include: plaque index, gingival index, probing depth, keratinized tissue, bleeding on probing, adjacent tooth recession, radiographic examination, tissue esthetics, colors, contours, and clinical photographs will be taken at baseline, during surgery and post-op visits.

The treatment will be randomly assigned using a coin toss. The mentor will flip the coin. The surgical procedure will consist of the reflection of full thickness flaps to expose the buccal crest. A dental implant will be placed in the edentulous site. Any implant system will be acceptable since the objective of the study is to evaluate soft tissue thickness and contour, not the dental implant. Either one layer of ADM or one layer of ADM plus bovine-derived xenograft (BX) will be placed following implant placement on the buccal aspect of the implant. When one layer of ADM is used it will be placed on the buccal surface of the implant only. When one layer of ADM and BX are used the BX will be overlaid buccal to the implant, then covered by ADM. Thus the buccal surface will have either one layer of ADM or one layer of ADM with BX. The surgical procedures will be documented with clinical photographs. Records will be kept of healing every 2 weeks for the first 8 weeks, then at 4 months or 16 weeks. At the end of 16 weeks or 4 months, once the study is completed, post and crown procedure over the implant can be started.

To provide adequate room to establish emergence profile the implant platform should be 3 to 4 mm apical to the mid-facial gingival margin when a 2-stage dental implant system is used. This may require reduction of the osseous crest by scalloping the bone so that the mid-facial osseous crest is 3-4 mm apical to the mid-facial gingival margin. This may result in a sub-crestal position of the interproximal implant platform (measured as a negative number). The top of the implant will be even with the crestal bone. The implant used will be any dental implant. At the time of surgery the implant platform will be placed even with the mid-facial osseous crest if a two-stage implant is used.

All probing measurements will be taken using the University of North Carolina probe. One investigator who is unaware of group assignment will perform all baseline examinations and all follow-up examinations. He will be calibrated prior to study initiation to assure that evaluations are consistent. The surgeon will perform all surgical procedures and will know the group to which each participant has been assigned. Standardized periapical radiographs will be taken at implant placement and at the 4-month examinations.

All patients will be seen at 1-2, 3-4, 5-6 and 7-8, and 16 weeks and buccal, occlusal and lingual clinical photographs will be taken at each visit. Patients will take doxycycline hyclate 100 mg qd for two weeks, Vicodin ES q4-6h as needed for pain, and naproxen 375 mg q12h for one week for inflammation. At post-operative visits plaque removal, and oral hygiene instruction, as needed, will be performed along with clinical photographs and standardized radiographs as scheduled.

ELIGIBILITY:
Inclusion Criteria:

1. Have one edentulous site bordered by 2 teeth in maxillary sites from second premolar to second premolar (maxillary 4 to 13) to receive an implant with simultaneous grafting with an ADM with or without bovine-derived xenograft.
2. Healthy persons at least 18 years old.
3. Understands and has signed the informed consent.

Exclusion Criteria:

1. Patients with uncontrolled diabetes, immune disease, or any systemic disease that significantly affects the periodontium.
2. Previous head and neck radiation.
3. Patients who have taken oral bisphosphonates for > 3 years or any IV bisphosphonates.
4. Smokers (or other tobacco habits that might interfere with soft tissue healing).
5. Patients who need prophylactic antibiotics prior to dental procedures.
6. Patients with allergies to any medication or material used in the study, or that would adversely affect study procedures.
7. Chemotherapy in the previous 12 months.
8. Psychological problems that would interfere with treatment.
9. Patients unable or unwilling to sign the informed consent.
10. Pregnant subjects will be excluded due to risk of miscarriage.

Post-treatment Exclusion Criteria

1. Failure of patient to follow treatment protocol.
2. Failure of implant to osseointegrate.
3. Failure of the allograft to heal.
4. Unanticipated healing complications that will adversely affect treatment results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Buccal soft tissue contour around dental implant. | 4 months post dental implant placement.
  Contour will be categorized as concave, flat, or convex (subjective categories).

SECONDARY OUTCOMES:
Buccal soft tissue thickness around dental implant. | 4 months post dental implant placement.
  Thickness will be measured with an endodontic file using a rubber stopper (objective measure of tissue thickness by penetrating tissue and measuring the thickness in mm).
Buccal soft tissue healing around dental implant. | 4 months post dental implant placement.
  The outcomes will be categorized as normal, delayed or accelerated (subjective assessment and assignment to a category).

CONTACTS AND LOCATIONS:
Overall Officials: Ting-wei H Hsu, D.M.D, Study Director — Co-investigator, University of Louisville; Henry Greenwell, D.M.D, M.S.D, Principal Investigator — University of Louisville; Bobby L Cockerham, DDS, Study Director — Co-investigator University of Louisville
Locations (1):
- Graduate Periodontics, University of Louisville School of Dentistry, Louisville, Kentucky, United States